CLINICAL TRIAL: NCT02482298
Title: A Randomised, Double-blind, Double-dummy, Parallel-group, Multicenter, Phase IIb Study to Evaluate the Effect of Ticagrelor Versus Placebo in Reducing the Number of Days With Pain in Young Adults With Sickle Cell Disease
Brief Title: A Study to Assess the Effect of Ticagrelor in Reducing the Number of Days With Pain in Patients With Sickle Cell Disease
Acronym: Hestia2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: D5136C00008
Record Dates: First submitted 2015-06-17; First posted 2015-06-26 (Estimated); Results first posted 2017-12-14 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease; Young adults; Hestia2; Ticagrelor
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dose A (Experimental)
  Interventions: Drug: Ticagrelor
- Dose B (Experimental)
  Interventions: Drug: Ticagrelor
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ticagrelor — Two arms: 1) 10 mg ticagrelor + 45 mg ticagrelor placebo or 2) 45 mg ticagrelor + 10 mg ticagrelor placebo. Drugs taken orally, twice a day (morning and evening, at least 12 hours apart) from randomization until the end of treatment.
  Arms: Dose A; Dose B
Drug: Placebo — 10 mg ticagrelor placebo + 45 mg ticagrelor placebo. Drugs taken orally, twice a day (morning and evening at least 12 hours apart) from randomization until the end of treatment
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether ticagrelor is effective in reducing the number of days of pain, intensity of pain, and reducing the use of analgesics due to sickle cell disease

DETAILED DESCRIPTION:
This is a randomised, double-blind, double-dummy, parallel-group, placebo-controlled, study evaluating 2 doses of ticagrelor in 90 patients aged 18 to 30 years, with sickle cell disease (SCD). Patients will be randomised to double-blind double-dummy treatment period in a 1:1:1 ratio (30 to each treatment group) to receive ticagrelor 10 mg twice daily (bid), or ticagrelor 45 mg bid, or placebo bid to determine the frequency of days with pain using an electronic diary (eDiary) every day. Approximately 180 patients will be enrolled. Patient will be followed for safety assessment during and after 2 weeks of treatment completion.

During the 16 week treatment period, patients will complete a daily eDiary concerning daily pain intensity, pain location, use of analgesics and absence from school or work. At the end of the study patients will be asked to rate the change in their sickle cell pain compared to the start of treatment. Platelet aggregation will be measured and reported as P2Y12 reaction units (PRU) pre-dose and 2 hours post-dose at week 4 and week 5 after treatment start. Pharmacokinetic (PK) parameters will be measured at 2 hours post-dose at week 4, and pre-dose and at 2 hours post-dose at week 5. Biomarkers will be assessed pre-dose at week 4, week 5 and week 8. During the study, patients will be evaluated for adverse events (AEs) including bleeding and vaso-occlusive crisis (VOC).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed medical history or diagnosis of homozygous sickle cell (HbSS) or sickle beta-zero-thalassaemia (HbS/β0) by HPLC
* If treated with hydroxyurea, the dose must have been stable for 3 months

Exclusion Criteria:

* History of transient ischaemic attack or clinically overt cerebrovascular accident
* Moderate or severe hepatic impairment
* Treatment with chronic red blood cell transfusion therapy
* Pre-dominate cause of pain is not sickle cell disease related
* Chronic treatment with anticoagulants or antiplatelet drugs.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2015-07-09 (Actual); Primary Completion 2016-11-16 (Actual); Study Completion 2016-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ignacia -Berraondo, MD, Study Director — Quintiles, Inc.
Locations (17):
- United States (3):
  - Research Site, Miami, Florida
  - Research Site, Bethesda, Maryland
  - Research Site, Charleston, South Carolina
- Egypt (2):
  - Research Site, Alexandria
  - Research Site, Cairo
- France (2):
  - Research Site, Bordeaux
  - Research Site, Strasbourg
- Research Site, Verona, Italy
- Kenya (3):
  - Research Site, Kikuyu
  - Research Site, Kisian
  - Research Site, Nairobi
- Research Site, Beirut, Lebanon
- Turkey (Türkiye) (3):
  - Research Site, Adana
  - Research Site, Mersin
  - Research Site, Van
- United Kingdom (2):
  - Research Site, Harrow
  - Research Site, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 26 centers in 8 countries between 09 July 2015 and 16 November 2016.
Pre-assignment Details: The study duration was approximately 18 weeks, consisting of a screening period including a 4-week single-blind placebo treatment for baseline assessments, a 12-week double-blind randomised treatment period, and a 2-week follow-up period. A total of 87 patients were randomized
Groups:
- TICAGRELOR 10MG BID + PLACEBO 45MG BID: Note that 1 patient in the Ticagrelor 10mg BID + Placebo 45mg BID group was excluded from the Safety analysis set because they had no post-dose assessments.
Period: Overall Study
Arm/Group | PLACEBO 10MG BID + PLACEBO 45MG BID | TICAGRELOR 10MG BID + PLACEBO 45MG BID | TICAGRELOR 45MG BID + PLACEBO 10MG BID
Started | 30 | 27 | 30
Completed | 28 | 24 | 27
Not Completed | 2 | 3 | 3
Not completed — Withdrawal by Subject | 2 | 1 | 2
Not completed — Did Not Fulfill Randomization Criteria | 0 | 1 | 0
Not completed — Dev. of Study-Spec. Withdrawal Criteria | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PLACEBO 10MG BID + PLACEBO 45MG BID | TICAGRELOR 10MG BID + PLACEBO 45MG BID | TICAGRELOR 45MG BID + PLACEBO 10MG BID | Total
Number analyzed (Participants) | 30 | 27 | 30 | 87
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.6 (3.42) [18 to 30] | 21.9 (2.72) [18 to 28] | 23.2 (3.69) [18 to 30] | 22.2 (3.35) [18 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 16 | 47
  Male | 14 | 12 | 14 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 15 | 14 | 17 | 46
  White | 15 | 12 | 13 | 40
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Proportion of Days With Pain Due to Sickle Cell Disease as Measured by an eDiary
Description: To investigate the efficacy of 2 different doses of ticagrelor versus placebo in reducing the number of days with pain due to sickle cell disease.
Time Frame: Baseline through Week 12
Population: The Efficacy analysis set included all randomized patients with at least 1 eDiary record post dose. Patients were analyzed according to their randomized IP.
Measure: Least Squares Mean (90% Confidence Interval); unit: Proportion of days with pain
Arm/Group | PLACEBO 10MG BID + PLACEBO 45MG BID | TICAGRELOR 10MG BID + PLACEBO 45MG BID | TICAGRELOR 45MG BID + PLACEBO 10MG BID
Number analyzed (Participants) | 30 | 27 | 30
Proportion of days with pain | -0.1802 (0.05453) [-0.2673 to -0.0931] | -0.1352 (0.05287) [-0.2260 to -0.0444] | -0.1001 (0.05233) [-0.1881 to -0.0121]
Statistical Analysis 1: Comparison: PLACEBO 10MG BID + PLACEBO 45MG BID vs TICAGRELOR 10MG BID + PLACEBO 45MG BID; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.0450, 90% CI 2-sided [-0.0610 to 0.1510], Standard Error of Mean 0.06367
Statistical Analysis 2: Comparison: PLACEBO 10MG BID + PLACEBO 45MG BID vs TICAGRELOR 45MG BID + PLACEBO 10MG BID; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.0801, 90% CI 2-sided [-0.0230 to 0.1832], Standard Error of Mean 0.06192

2. Secondary Outcome: Average of the Daily Worst Pain Values Reported Via eDiary
Description: To determine the efficacy of 2 different doses of ticagrelor versus placebo in reducing the intensity of pain due to sickle cell disease. Intensity of pain was recorded on an 11-point scale where 0 represented no pain and 10 represented the worst pain imaginable.
Time Frame: Baseline through Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Average daily worst pain rating
Arm/Group | PLACEBO 10MG BID + PLACEBO 45MG BID | TICAGRELOR 10MG BID + PLACEBO 45MG BID | TICAGRELOR 45MG BID + PLACEBO 10MG BID
Number analyzed (Participants) | 30 | 27 | 30
Average daily worst pain rating | 1.02 (1.106) | 1.15 (1.547) | 1.74 (2.277)

3. Secondary Outcome: Change in Proportion of Days With Analgesic Use Measured by an eDiary
Description: To assess the efficacy of 2 different doses of ticagrelor versus placebo in reducing the use of analgesics by patients with sickle cell disease.
Time Frame: Baseline through Week 12
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: Proportion of days with analgesic use
Arm/Group | PLACEBO 10MG BID + PLACEBO 45MG BID | TICAGRELOR 10MG BID + PLACEBO 45MG BID | TICAGRELOR 45MG BID + PLACEBO 10MG BID
Number analyzed (Participants) | 30 | 27 | 30
Proportion of days with analgesic use | -0.1991 (0.08763) [-0.2753 to -0.1230] | -0.0799 (0.08540) [-0.1590 to -0.0008] | -0.1016 (0.08664) [-0.1782 to -0.0250]
Statistical Analysis 1: Comparison: PLACEBO 10MG BID + PLACEBO 45MG BID vs TICAGRELOR 10MG BID + PLACEBO 45MG BID; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.1192, 90% CI 2-sided [0.0350 to 0.2035], Standard Error of Mean 0.05059
Statistical Analysis 2: Comparison: PLACEBO 10MG BID + PLACEBO 45MG BID vs TICAGRELOR 45MG BID + PLACEBO 10MG BID; Test type: Superiority or Other; Mixed Models Analysis; Mean Difference (Final Values) = 0.0975, 90% CI 2-sided [0.0155 to 0.1795], Standard Error of Mean 0.04923

4. Other Pre Specified Outcome: Number of Major Bleeding or Clinically Relevant Non-major Bleeding Events (Patients)
Description: To assess safety and tolerability of 2 different doses of ticagrelor versus placebo in patients with SCD
Time Frame: Baseline through Week 12
Population: The Safety analysis set included all patients who received at least 1 single dose of randomised IP, ticagrelor or placebo, and for whom any post-dose data were available. Patients were analysed according to the actual treatment.
Measure: Number; unit: Number of patients
Arm/Group | PLACEBO 10MG BID + PLACEBO 45MG BID | TICAGRELOR 10MG BID + PLACEBO 45MG BID | TICAGRELOR 45MG BID + PLACEBO 10MG BID
Number analyzed (Participants) | 30 | 26 | 30
Number of patients
  Patients with any bleeding events | 2 | 2 | 2
  Pts w/ any bleeding event requiring intervention | 2 | 1 | 2

5. Other Pre Specified Outcome: Number of Major Bleeding or Clinically Relevant Non-major Bleeding Events (Events)
Description: To assess safety and tolerability of 2 different doses of ticagrelor versus placebo in patients with SCD
Time Frame: Baseline through Week 12
Population: as for outcome 4
Measure: Number; unit: Number of events
Arm/Group | PLACEBO 10MG BID + PLACEBO 45MG BID | TICAGRELOR 10MG BID + PLACEBO 45MG BID | TICAGRELOR 45MG BID + PLACEBO 10MG BID
Number analyzed (Participants) | 30 | 26 | 30
Number of events
  Total number of bleeding events | 2 | 2 | 2
  Maximum severity of bleeding event: Minor | 0 | 1 | 0
  Max sever. of bleed event: Clin-relevant nonmajor | 2 | 1 | 2
  Maximum severity of bleeding event: Major | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | PLACEBO 10MG BID + PLACEBO 45MG BID | TICAGRELOR 10MG BID + PLACEBO 45MG BID | TICAGRELOR 45MG BID + PLACEBO 10MG BID
Serious Adverse Events (participants affected / at risk) | 6/30 | 6/26 | 5/30
Other Adverse Events (participants affected / at risk) | 16/30 | 15/26 | 20/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO 10MG BID + PLACEBO 45MG BID (N=30) | TICAGRELOR 10MG BID + PLACEBO 45MG BID (N=26) | TICAGRELOR 45MG BID + PLACEBO 10MG BID (N=30)
Reticulocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 3 (7) | 5 (6) | 3 (3)
Local swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic ischaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vascular occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO 10MG BID + PLACEBO 45MG BID (N=30) | TICAGRELOR 10MG BID + PLACEBO 45MG BID (N=26) | TICAGRELOR 45MG BID + PLACEBO 10MG BID (N=30)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 (3) | 1 (1) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 5 (11) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (3) | 2 (2)
Fatigue (General disorders) | 2 (2) | 1 (1) | 2 (2)
Non-cardiac chest pain (General disorders) | 3 (4) | 3 (10) | 4 (10)
Pain (General disorders) | 1 (1) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 2 (4) | 2 (2) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (5) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (23) | 6 (21) | 9 (47)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (20) | 4 (10) | 4 (12)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (7)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (5) | 3 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (11) | 4 (12) | 9 (22)
Headache (Nervous system disorders) | 8 (23) | 11 (25) | 8 (28)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Public disclosure of trial results by Principle Investigators within two years of trial completion requires Sponsor's prior written consent.